CLINICAL TRIAL: NCT05821491
Title: Prognosis of Geriatric Patients With Non-bedded Night in the Emergency Department: a Multicenter Cohort Study
Acronym: NoBedNight
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221326
Record Dates: First submitted 2022-12-16; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: in Hospital Mortality; Geriatric
Keywords: In-hospital mortality; Geriatric patient; Emergency unit; No-bedding night
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-bedded night: geriatric patients with non-bedded night in the emergency department
- bedded night: geriatric patients with bedded night in the emergency department

SUMMARY:
Retrospective, multicenter, French cohort study. Data from patients over 75 years of age who visited the emergency department on 12 and 13 December 2022 could be collected until their discharge from hospital and for a maximum of 30 days. Data from patients who spent the night on a stretcher (stretcher group) as well as from a group of patients who spent the night in a bed (hospital bed group) after a visit to the emergency department will be collected.

The characteristics of the patients and their stay in the emergency room will be collected, and their hospital stay (truncated at 30 days) will be analyzed in terms of morbidity and mortality.

Main objective:

To study the truncated 30-day in-hospital mortality of patients who spent a night on a stretcher in the emergency department.

Secondary objectives:

To describe the characteristics and hospital stay of patients who spent a night on a stretcher To compare the morbidity and mortality of patients who spent the night on a stretcher with patients who spent the night in an inpatient bed after an emergency visit;

DETAILED DESCRIPTION:
The activity and number of admissions to emergency departments are constantly increasing, resulting in the overloading of emergency departments, a problem shared by most Western countries, for a variety of reasons. The ageing of the population and the increasing scarcity of outpatient medical services have led to an increase in the number of consultations in emergency departments by patients aged over 75. These demographic changes and the reduction in the number of hospital beds in France have led to overcrowding in emergency departments (EDs), with long waiting times for patients to be admitted to hospital. Emergency department overcrowding is directly associated with an increase in mortality at 24 hours (adjusted OR 1.42; 95%CI 1.08-1.88) and at 72 hours (adjusted OR 1.27; 95%CI 1.02-1.58) after a visit to the emergency department. Similarly, several retrospective studies report an association between in-hospital mortality and the time spent in the emergency department, and the time spent waiting for a hospital bed in particular.

The No Bed Challenge, organised by Samu Urgences de France (SUDF) in 2018, identified patients who spent the night on a stretcher waiting for a hospital bed. Beyond the long waiting time and its association with excess mortality, spending the night on a stretcher can be associated with a worsening prognosis: the conditions of care and comfort are degraded, and the risks inherent in such a nightly wait on a stretcher are multiple. It has been described that beyond 5 hours, waiting is linked with a linear increase in 30-day mortality. In addition, several retrospective studies report a longer waiting time for a downstream hospitalization bed for the geriatric patient population. This longer waiting time is also associated with the occurrence of adverse events, increasing by 3% for each hour spent in the emergency department. However, the characteristics of patients spending the night in the emergency department while waiting for a hospital bed, and their prognosis, are not known - particularly in France.

The objective of the NoBedNight study is to study the in-hospital mortality of patients over 75 years old who spent the night on a stretcher. It will also allow us to describe the typology of these patients, and to compare them to a similar population who had access to an outpatient bed after a visit to the emergency room.

The study aim to evaluate the in-hospital mortality of patients over 75 years old spending the night on a stretcher in the emergency room while waiting for an inpatient bed by collecting data collected in the course of care.

This national retrospective multicentre cohort study will provide information on the clinical characteristics of this population, their frailty index (assessed by Charlson's Comorbidity Index) and their level of dependence (GIR scale) which will be calculated a posteriori on the data collected during care, as well as their clinical presentation, their reason for referral and the occurrence of complications during hospitalisation.

It will make it possible to evaluate the number of geriatric patients waiting for a hospital bed over a short-predefined period in our French emergency services.

The increase in the overload of emergency departments leads to regular national crises in France and in Western countries. It is important to assess the consequences on the health of patients, particularly geriatric patients.

According to the literature, the hypothesis is that mortality is increased in geriatric patients who spend a night on a stretcher in an emergency department because they do not have an inpatient bed.

In recent years, many ideas have been put forward to alleviate the overloading of emergency departments, the cause of which is multifactorial. However, obtaining precise and updated data will make it possible to evaluate the magnitude of the risks inherent in waiting for an outpatient hospital bed for elderly patients and to conclude on the mortality of patients at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 75 years of age
* Emergency department patient between 12 December 8am and 14 December 8am.
* Having spent the whole of one of the 2 periods midnight-8am on a stretcher in the ED ("stretcher" group), or in an inpatient bed (including short hospitalization unit) ("inpatient bed" group).

Decision to hospitalise after discharge from the emergency department (excluding the continuous care unit)

Exclusion Criteria:

* Patient admitted to an inpatient bed between midnight and 8am
* Patient discharged home

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All data of eligible patients over 75 years old who visited the emergency departments of the concerned hospitals on 12 and 13 December 2022 will be collected.
  These data will be broken down into :
  * Patients who spent the night on a stretcher,
  * Patients who spent the night in a bed after an emergency visit.
Sampling Method: Non-Probability Sample
Enrollment: 1598 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | 30 days after ED's admission
  To study in-hospital mortality, truncated at 30 days, of patients who spent a night on a stretcher in the emergency department

SECONDARY OUTCOMES:
Lenght of hospital stay in days | End of hospitalization, truncated at 30 days
  Describe the hospital stay of patients who spent a night on a stretcher
Morbidity | End of hospitalization, truncated at 30 days
  To compare the morbidity (complications arising during hospitalisation) of these patients who did not spend the night on a stretcher with those who spent the night in an inpatient bed after an emergency visit

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No